CLINICAL TRIAL: NCT01802463
Title: Correlation Between Ocular Blood Flow and the Optic Nerve Sheath Diameter in Patients With Primary Open-angle Glaucoma
Brief Title: Study on Ocular Blood Flow and the Orbital Cerebrospinal Fluid Pressure in Glaucoma
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S130213
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-01

CONDITIONS: Open Angle Glaucoma; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls: Healthy volunteers with no family history of glaucoma, an increased or asymmetrical cup/disc ratio or any other optic disc structural change (notching, disc hemorrhage) or an intraocular pressure (IOP) above 21 mmHg that could suggest possible glaucoma suspects.
- Primary open-angle glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at least one measurement of IOP of >21 mmHg required
- Normal Tension Glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at maximum recorded IOP of < 21 mmHg

SUMMARY:
Ocular blood flow has been consistently demonstrated to be altered in glaucoma patients when compared to otherwise healthy individuals. Numerous Doppler studies have shown a decrease in flow velocities in the retrobulbar arteries in what appears to be related to the degree of the glaucomatous disease.

The anatomic pathway of the several arteries into the eye is intricately complicate, with at least one of them (the central retina artery) penetrating the optic nerve before entering the eye and supplying the innermost structures of the globe. As the optic nerve is surrounded by a layer of cerebrospinal fluid (CSF) which is in continuity with the rest of the central nervous system, this central retinal artery has also to cross this CSF containing compartment. Because of the intrinsic pressure this CSF - corresponding to the intracranial pressure at the orbital level - the possibility exists that this pressure around the optic disc could affect the blood flow of the arteries that go through it.

The investigators will try to detect if a correlation exists between the optic nerve sheath diameter and the blood flow in the retrobulbar vessels of glaucoma patients.

DETAILED DESCRIPTION:
1. Visual field testing will be performed.
2. Structural analysis of the retinal nerve fiber layer (through confocal microscopy)will be performed.
3. Color Doppler Imaging of the retrobulbar vessels will be performed. Peak and end diastolic velocities, resistivity index will be calculated from the Doppler waveform.
4. B-scan ultrasound of the optic nerve sheath diameter will be performed. the measure will take place at 3mm behind the globe.

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply with the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for cataract surgery)
* eye disease (except glaucoma)
* systemic diseases with ocular involvement like diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary clinic care
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Flow velocity of retrobulbar vessels | Participants will be followed for the duration of hospital stay, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Flemish Brabant, Belgium

REFERENCES:
- [Derived] Willekens K, Abegao Pinto L, Vandewalle E, Marques-Neves C, Stalmans I. Higher optic nerve sheath diameters are associated with lower ocular blood flow velocities in glaucoma patients. Graefes Arch Clin Exp Ophthalmol. 2014 Mar;252(3):477-83. doi: 10.1007/s00417-013-2533-y. Epub 2013 Nov 27. PMID 24281785